CLINICAL TRIAL: NCT01544023
Title: Multicenter Observational Study of Implant Based Breast Reconstruction Using a Titanium-coated Polypropylene Mesh
Brief Title: TiLoop® Bra for Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Max Dieterich, Principle investigator, University of Rostock
Other Study IDs: TL001
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2016-12

CONDITIONS: Patient and Surgical Related Risk Factors for Complications
Keywords: breast reconstruction; mesh; implant reconstruction; acellular dermal matrix; titanized polypropylene mesh; TiLOOP Bra; TiLOOP; implant based breast reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Reconstruction with TilOOP

SUMMARY:
A new approach for single stage implant based breast reconstruction (BR) is the use of a titanium-coated polypropylene mesh (TCPM) as an alternative to acellular dermal matrix (ADM). These TCPM have a good biocompatibility and can be used in a similar way as ADM. This study addresses indications, limitations and complications of TCPM in implant based breast reconstruction.

DETAILED DESCRIPTION:
An alternative to ADM is the usage of a titanium-coated polypropylene mesh (TCPM=TiLOOP(R) Bra), which is approved for breast reconstruction in Europe. The surgical approach is identical in comparison to ADM reconstruction and has been described previously. This titanium coated lightweight mesh consists of a monofilament structure and was initially invented for hernia repair which has a good biocompatibility. Observed cellular reactions like proliferation and apoptosis were at the lowest level when using this lightweight TCPM compared to not titanium-coated meshes (pure polypropylene (PP), pure lightweight PP mesh or PP mesh incorporating resorbable polyglactic acid). Histopathological analysis of an intraoperative sample of a TCPM after expander/implant BR demonstrated a well incorporated mesh with only weak inflammatory reactions. Preliminary data of in-vitro investigations at the investigators institute confirms the good biocompatibility of this TCPM in distinctive breast tissues (fibroblasts, fat cells, muscle cells) Although meshes are used in a large scale there are no sufficient clinical data regarding safety and outcome. In this multicenter study the investigators are able to investigate a large cohort of patients undergoing implant based breast reconstruction using a TCPM.

ELIGIBILITY:
Inclusion Criteria:

* Indication for immediate or secondary implant based breast reconstruction

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for immediate or secondary implant based breast reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max Dieterich, MD, Principal Investigator — University of Rostock; Bernd Gerber, Prof., Study Chair — University of Rostock

REFERENCES:
- [Derived] Dieterich M, Paepke S, Zwiefel K, Dieterich H, Blohmer J, Faridi A, Klein E, Gerber B, Nestle-Kraemling C. Implant-based breast reconstruction using a titanium-coated polypropylene mesh (TiLOOP Bra): a multicenter study of 231 cases. Plast Reconstr Surg. 2013 Jul;132(1):8e-19e. doi: 10.1097/PRS.0b013e318290f8a0. PMID 23806958

RESULTS

PARTICIPANT FLOW:
Groups:
- TiLOOP: Patients with immediate or delayed-immediate heterologous BR who underwent skin-sparing (SSM) or nipple-sparing mastectomy (NSM) with silicone implants in combination with TiLOOP" Bra (pfm medical, Cologne, Germany) were included.
Period: Overall Study
Arm/Group | TiLOOP
Started | 207 (retrospective)
Completed | 207
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TiLOOP
Number analyzed (Participants) | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (11.6)
Gender [Count of Participants; unit: Participants]
  Female | 207
  Male | 0
Region of Enrollment [Number; unit: participants]
  Germany | 207

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Received TiLOOP Mesh Reconstruction
Description: Primary study endpoint was the identification of patient- and surgical factors predictive of adverse outcome and to develop recommendations for patients eligible for implant based breast reconstruction (IBBR) using TCPM.
Time Frame: 1 month
Measure: Number; unit: Patients with TiLOOP mesh reconstruction
Arm/Group | TiLOOP
Number analyzed (Participants) | 207
Patients with TiLOOP mesh reconstruction | 207

2. Secondary Outcome: Complication Rate
Description: Secondary study outcome was the prevalence of complications.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | TiLOOP
Number analyzed (Participants) | 207
percentage of participants
  Major Complications | 13.4
  Minor Complications | 15.6

ADVERSE EVENTS:
Time Frame: Retrospective chart analysis. With Follow up up to 2 years
Description: Adverse Events were not collected/assessed.
Arm/Group | TiLOOP
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes